CLINICAL TRIAL: NCT00874575
Title: A Double Blind Study on the Efficacy of a Combination of Beta-hydroxy-beta-methylbutyrate and Vitamin D on Muscular Strength and Functionality in Older Adults.
Brief Title: Nutritional Intervention for Age-related Muscular Function and Strength Losses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: Iowa State University (Other); South Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: MTI2008-CS01
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Muscle Strength; Sarcopenia
Keywords: HMB; Vitamin D; Older Adults
MeSH Terms: conditions — Sarcopenia | interventions — Vitamin D; Cholecalciferol; beta-hydroxyisovaleric acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Control
  Interventions: Dietary Supplement: Placebo
- 2 (Experimental): Beta-hydroxy-Beta-methylbutyrate, 3 g/d
  Interventions: Dietary Supplement: Beta-hydroxy-Beta-methylbutyrate
- 3 (Experimental): Vitamin D, 2000 IU/d
  Interventions: Dietary Supplement: Vitamin D
- 4 (Experimental): Beta-hydroxy-Beta-methylbutyrate (3 g/d) + Vitamin D (2000 IU/d)
  Interventions: Drug: Beta-hydroxy-Beta-methylbutyrate and Vitamin D

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: 1
Dietary Supplement: Vitamin D
  Other Names: Cholecalciferol
  Arms: 3
Dietary Supplement: Beta-hydroxy-Beta-methylbutyrate
  Other Names: HMB
  Arms: 2
Drug: Beta-hydroxy-Beta-methylbutyrate and Vitamin D
  Other Names: Beta-hydroxy-Beta-methylbutyrate: HMB; Vitamin D: Cholecalciferol
  Arms: 4

SUMMARY:
The purpose of the study is to

* Test the effect of a dietary supplement beta-hydroxy-beta-methylbutyrate (HMB) with and without Vitamin D to prevent and reverse the losses of muscular strength and functionality in older adults.

The second aim of the study is to determine if HMB and Vitamin D improves markers of bone turnover in adults aged 60 plus years. HMB is a dietary supplement that comes from the amino acid leucine. HMB is found in foods and is made in your body after you eat protein (meat). Subjects will be randomized to one of four dietary supplement groups and will participate in a 3-day per week exercise program for 12 weeks. Each exercise day will be about 60 minutes long consisting of strength training exercises utilizing Theraband® stretch cords and jumping.

Subjects will consume the dietary supplement 2 times per day for 12 weeks. Tests will consist of the following:

* Measuring the strength of subjects' legs by using a Isokinetic Dynamometer
* Measuring body composition
* Measuring hand-grip strength using a hand-grip dynamometer
* Measuring functional mobility, balance and agility by the time it takes for you to rise from a chair, walk around a cone 8 feet in front of the chair and return to the chair (Up-&-Go Test
* Filling out questionnaires and having blood drawn for biochemical measurements. Testing will be performed at the beginning and at 4, 8 and 12 weeks.

ELIGIBILITY:
Subjects must meet all of the inclusion criteria in order to participate in the study.

* Male and Female subjects will be enrolled into the study.
* Age > 60 years.
* Free of liver and kidney diseases, and with no evidence of uncontrolled hypertension.
* Does not have a chronic disease that affects calcium or bone metabolism (i.e., asthma with chronic use of high dose steroids, inflammatory bowel disease, Crohn's disease, primary hyperparathyroidism, seizure disorder with use of phenobarbital, etc.).
* Not classified as morbidly obese (body mass index (BMI) >40 kg/m2).
* Six weeks since major surgery (three weeks since minor surgery).
* Willing to consume one of the nutritional supplements for the study period.
* Individuals diagnosed with osteoporosis (i.e., bone density > 2.5 standard deviations below the mean) will not be enrolled in the study.
* No other serious medical illness.
* Serum 25OH-VitD3 >10 and <25 ng/ml.
* Able and willing to participate in 3-day-a-week monitored strength-training program.
* Physician has placed no restriction on physical exercise.

All candidates meeting any one of the exclusion criteria will not be enrolled into the study and as necessary will be referred to their private physician for further follow-up.

* Age < 60 years.
* Evidence of liver and kidney diseases, uncontrolled hypertension, or Type I diabetes mellitus requiring insulin for glucose control.
* Presence of a chronic disease that affects calcium or bone metabolism (i.e., asthma with chronic use of high dose steroids, inflammatory bowel disease, Crohn's disease, primary hyperparathyroidism, seizure disorder with use of phenobarbital, etc.).
* Classified as morbidly obese (body mass index (BMI) >40 kg/m2).
* Less than six weeks since major surgery or three weeks since minor surgery.
* Not willing to consume one of the nutritional supplements for the study period.
* Individuals diagnosed with osteoporosis (i.e., bone density > 2.5 standard deviations below the mean) will not be enrolled in the study.
* Other serious medical illness, which the subjects doctor or medical review team has decided affects the subject's ability to participate in the study.
* Subjects on high dose vitamin D therapies (i.e. 50,000 IU vitamin D).
* Subjects with serum 25OH-VitD3 <10 ng/ml will be considered deficient and will be referred to their physician for treatment.
* Subjects with serum 25OH-VitD3 >25 ng/ml.
* Not able or willing to participate in 3-day-a-week monitored strength-training program.
* Physician has placed a restriction on physical exercise.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Muscular Strength and functionality | 12 weeks

SECONDARY OUTCOMES:
Bone turnover | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John A. Rathmacher, Ph.D., Principal Investigator — Metabolic Technologies
Locations (2):
- United States (2):
  - Iowa State University, Ames, Iowa
  - South Dakota State University, Brookings, South Dakota